CLINICAL TRIAL: NCT01033253
Title: Multi-media Obesity Prevention Program for Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pro-Change Behavior Systems (Other)
Responsible Party: Leanne Mauriello, Pro-Change Behavior Systems, Inc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R44HL074482-02 (NIH)
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2009-12

CONDITIONS: Physical Activity; Nutrition; Obesity Prevention
MeSH Terms: conditions — Motor Activity | interventions — Health; Motion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computerized Tailored Intervention (Experimental): Students interacted with the 30-minute program through a series of Transtheoretical Model (TTM) based assessments and tailored feedback messages. A full TTM intervention was delivered for physical activity, in which each of the appropriate constructs of the TTM based on stage of change was addressed. Optimally tailored interventions were delivered for fruit and vegetable consumption and limited TV viewing. These interventions offered feedback on the most important TTM constructs based on stage of change for each behavior. Multimedia components, including audio, video, and animations helped to capture students' interest.
  Interventions: Behavioral: Health in Motion
- Control (No Intervention): Computerized assessments of Transtheoretical Model constructs at 0, 2, 6, and 12 months

INTERVENTIONS:
Behavioral: Health in Motion — Students interacted with the 30-minute program through a series of Transtheoretical Model (TTM) based assessments and tailored feedback messages. A full TTM intervention was delivered for physical activity, in which each of the appropriate constructs of the TTM based on stage of change was addressed. Optimally tailored interventions were delivered for fruit and vegetable consumption and limited TV viewing. These interventions offered feedback on the most important TTM constructs based on stage of change for each behavior. Multimedia components, including audio, video, and animations helped to capture students' interest.
  Arms: Computerized Tailored Intervention

SUMMARY:
The objective of this project was to evaluate a population-based, computerized tailored intervention that addresses recommended guidelines for three target behaviors related to obesity risk: physical activity (at least 60 minutes on at least 5 days per week), fruit and vegetable consumption (at least 5 servings of fruits and vegetables each day), and limited TV viewing (2 hours or less of TV each day).

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* In the 9th, 10th, or 11th grade at baseline

Exclusion Criteria:

-

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1800 (Actual)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The number of days per week for which students got at least 60 minutes of physical activity | 2, 6, and 12 months
The number of servings of fruits and vegetables consumed each day | 2, 6, and 12 months
The number of hours of TV watch each day, including time spent watching TV, videotapes, and DVD's | 2, 6, and 12 months

SECONDARY OUTCOMES:
Stage of change for readiness to do at least 60 minutes of physical activity on at least 5 days of the week | 2, 6, and 12 months
Stage of change for readiness to eat at least five servings of fruits and vegetables each day. | 2, 6, and 12 months
Stage of change for readiness to watch two hours or less of TV each day. | 2, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Mauriello, Ph.D., Principal Investigator — Pro-Change Behavior Systems
Locations (1):
- Pro-Change Behavior Systems, Inc., Kingston, Rhode Island, United States

REFERENCES:
- [Background] Driskell MM, Dyment S, Mauriello L, Castle P, Sherman K. Relationships among multiple behaviors for childhood and adolescent obesity prevention. Prev Med. 2008 Mar;46(3):209-15. doi: 10.1016/j.ypmed.2007.07.028. Epub 2007 Aug 1. PMID 17714771
- [Background] Mauriello LM, Driskell MM, Sherman KJ, Johnson SS, Prochaska JM, Prochaska JO. Acceptability of a school-based intervention for the prevention of adolescent obesity. J Sch Nurs. 2006 Oct;22(5):269-77. doi: 10.1177/10598405060220050501. PMID 17172199
- [Background] Mauriello LM, Sherman KJ, Driskell MM, Prochaska JM. Using interactive behavior change technology to intervene on physical activity and nutrition with adolescents. Adolesc Med State Art Rev. 2007 Aug;18(2):383-99, xiii. PMID 18605653